CLINICAL TRIAL: NCT05031923
Title: Treatment of Intrabony Defects With Simvastatin and Antimicrobial Photodynamic Therapy: A Randomized Controlled Clinical Trial
Brief Title: Treatment of Intrabony Defects With Simvastatin and Antimicrobial Photodynamic Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, Principle investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: waiting..
Record Dates: First submitted 2021-08-20; First posted 2021-09-02 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Simvastatin; Photodynamic Therapy; Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMV and antimicrobial photodynamic therapy (Experimental): Application SMV and antimicrobial photodynamic therapy in intrabony defect
  Interventions: Procedure: SMV and antimicrobial photodynamic therapy
- SMV application (Active Comparator): Application SMV in intrabony defect
  Interventions: Procedure: SMV application

INTERVENTIONS:
Procedure: SMV and antimicrobial photodynamic therapy — Application of SMV and antimicrobial photodynamic therapy in intrabony defects
  Arms: SMV and antimicrobial photodynamic therapy
Procedure: SMV application — Application of SMV without antimicrobial photodynamic therapy in intrabony defects
  Arms: SMV application

SUMMARY:
Antimicrobial photodynamic therapy (aPDT) is characterized by the association of photosensitizing agents, promoting the generation of reactive oxygen species like free radicals and singlet oxygen, which are cytotoxic to certain bacteria. Simvastatin (SMV) enhances alkaline phosphatase activity and increases the expression of bone sialoprotein, osteocalcin, and type I collagen and is shown to have an anti-inflammatory effect by decreasing the production of C-reactive protein (CRP), IL-6, and IL-8. SMV is also reported to stimulate VEGF release in a dose-dependent manner which promotes osteoblast differentiation and bone nodule formation. The aim of this study is to evaluate the adjunctive effects of SMV with and without aPDT in chronic periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients were all healthy and free from any systemic disease;
* no history of antibiotic therapy or periodontal treatment for at least 6 months preceding the study;
* patients were willing and able to return for multiple follow-up visits;
* good levels of oral hygiene

Exclusion Criteria:

* Pregnant and lactating female patients,
* smokers,
* alcoholics,
* those receiving any medication that could affect healing of soft or hard tissue

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-16 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation and measurements of the defect in millimeters | 9 months
  Changes in clinical measurements after application of simvastatin with and without antimicrobial photodynamic therapy in millimeters
Radiographic evaluation and measurements of the defect in millimeters | 9 months
  Changes in bone formation in millimeters after application of simvastatin with and without antimicrobial photodynamic therapy in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Egypt